CLINICAL TRIAL: NCT06563622
Title: Ultrasound-Guided Pericapsular Nerve Group Block Versus Ultrasound-Guided Caudal Block for Postoperative Pain Management in Pediatric Hip Surgery; a Randomized Controlled Trail
Brief Title: Pericapsular Nerve Group Block Versus Caudal Block for Postoperative Pain Management in Pediatric Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, Assistant professor of anaesthesia and intensive care, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC.30.9.2023
Record Dates: First submitted 2024-08-13; First posted 2024-08-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Experimental): In ultrasound-guided pericapsular nerve group block Group , the patient will be positioned in a supine position. The anatomical landmarks, including ilio-pubic eminence, the iliopsoas muscle and tendon, the femoral artery and vein, and the pectineus muscle, will be identified using a 9-12 MHz superficial linear transducer. A lateral to medial in-plane technique will be used to insert a 22-gauge, 50-mm needle. the needle's tip will be positioned at the musculofascial plane, located between the ilio-pubic ramus posteriorly and the psoas tendon anteriorly. Following negative aspiration to avoid intravascular injection, 0.5-1 ml of normal saline will be injected to confirm the correct needle site. A 0.5 ml/kg plain bupivacaine 0.25% will be injected.
  Interventions: Procedure: Pericapsular Nerves Group Block
- Group C (Active Comparator): the caudal epidural block will be established in the lateral decubitus position, the high-frequency linear transducer will be first placed transversely at the midline to obtain a "frog eye" sign view of the sacral cornu, the sacro-coccygeal ligament, the sacrum, and the sacral hiatus. At this position, the USG transducer will be rotated by 90° to obtain a longitudinal view. The needle will be inserted in-plane into the sacral canal and the Local anaesthetics will be injected under real-time visualization by a dose of 0.5 ml/kg plain bupivacaine 0.25%.
  Interventions: Procedure: Caudal Epidural Block

INTERVENTIONS:
Procedure: Pericapsular Nerves Group Block — USG-guided single-shot PENG in a dose of 0.5 ml/kg of 0.25% bupivacaine per side.
  Other Names: PENG Block
  Arms: Group P
Procedure: Caudal Epidural Block — USG-guided single-shot CEB in a dose of 0.5 mL/kg of 0.25% bupivacaine.
  Other Names: CEB
  Arms: Group C

SUMMARY:
Children can experience substantial pain after hip operations, causing agitation, depression, and sleep disruption, which can have a negative impact on their health. Opioids are associated with several serious side effects that limits its use as solo agents for pain management. Regional blocks such as caudal Block (CB) and pericapsular nerve group (PENG) block in adjuvant with general anaesthesia are alternative perioperative analgesic techniques that lead to lesser side effects, including motor weakness, postoperative nausea and vomiting with decreased opioid consumption.

DETAILED DESCRIPTION:
Regional anesthesia is often used to prevent postoperative pain in pediatric surgery. Combined with general anesthesia (GA), ultrasound (US)-guided regional anesthetic approaches provide simple intraoperative pathway that reduced GA requirements, lower pain score with less impact on the respiratory or cardiovascular system

In pediatric surgery, caudal block (CB) is a low-cost, simple, and effective procedure for postoperative analgesia. CB is suggested for most surgeries in the lower body, primarily below the umbilicus. Although the well-established anesthetic properties of CB, its action terminates early in the postoperative period and it has a number of restrictions, such as anatomical abnormalities or infection at the injection site, that can prevent its use

PENG block is the plane lying between the psoas muscle and tendon and the ilio-pubic eminence. The single-shot PENG block has lately been reported in the cadaveric study and in the literature for perioperative pain management in hip surgery by aiming the articular arms of the accessory obturator nerve (AON), femoral nerve (FN), and obturator nerve (ON). The technical simplicity of imaging in traction-fixed patients and no need for multiple punctures made this blockage ideal for young pediatric patients. Unfortunately, there are no adequate studies regarding PENG block in patients younger than five years old.

This study was carried out to assess ultrasound-guided PENG block versus CB for their efficacy, safety and pain management in pediatric hip surgery.

ELIGIBILITY:
Inclusion Criteria:

* child aged 1- 7 years old
* American Society of Anesthesiologists (ASA) physical status I-II
* scheduled for elective hip surgery under general anesthesia

Exclusion Criteria:

* parents/guardians refusal to participate
* known local anesthetic drug sensitivity,
* bleeding disorders,
* pre-existing infection at the block site, and
* the presence of major cardiac, renal, or hepatic disorders.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
pain score with FLACC | 30 minutes postoperative, 1 hour postoperative, 2 hour postoperative, and 6 hours postoperative
  (Face, Legs, Activity, Cry, and Consolability scale to assess pain in young children. Each category is scored on a 0-2 scale which results in a total score between 0 (lowest pain) and 10 (worst pain).

SECONDARY OUTCOMES:
The duration of the block | immediately after the intervention, up to 24 hours postoperative
  from immediately after the block administration until the first postoperative rescue analgesia.
the Time to first postoperative rescue analgesia | 24 hours postoperative
  it will be administered if the FLACC score is ≥ 4/10.
Total rescue analgesia consumption | 24 hours postoperative
  total dose of Morphine administrated as rescue opioid
The incidence of postoperative adverse effects | 24 hours postoperative
  including nausea , vomiting , localized hematoma, bradycardia, hypo-tension, and Pruritis.
Parents satisfaction score | 24 hours postoperative
  using a 5- point Likert score (0 = very dissatisfied, 1=dissatisfied, 2 = neither satisfied nor dissatisfied, 3 = satisfied and 4 = very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Rafik Mohamed Amin, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No